CLINICAL TRIAL: NCT03821883
Title: Aspirin Discontinuation After Left Atrial Appendage Occlusion in Atrial Fibrillation
Acronym: ASPIRIN-LAAO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XH-18-017
Record Dates: First submitted 2019-01-22; First posted 2019-01-30 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-06

CONDITIONS: Atrial Fibrillation; Stroke; Bleeding
Keywords: Atrial fibrillation; Stroke; Left atrial appendage closure; Aspirin
MeSH Terms: conditions — Atrial Fibrillation; Stroke; Hemorrhage | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aspirin group (Experimental): Study patients assigned to Aspirin group will receive enteric coated aspirin (100 mg/day).
  Interventions: Drug: Aspirin Tablet
- Control group (Placebo Comparator): Study patients assigned to control group will receive placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aspirin Tablet — Aspirin 100mg qd
  Arms: Aspirin group
Drug: Placebo — Placebo qd
  Arms: Control group

SUMMARY:
The ASPIRIN LAAO trial is a prospective, multi-center, randomized, double blinded, placebo-controlled study aiming at investigating the safety of terminating the use of aspirin after left atrial appendage occlusion (LAAO).

Patients diagnosed with atrial fibrillation and have undergone LAAO will be enrolled in this study. Randomization will be performed at 6 months post-implant. The randomization program electronically assigns the patient 1:1 to either the Aspirin group or the control group. Study patients assigned to Aspirin group will receive enteric coated aspirin (100 mg/day). The control group receives placebo. After the randomization, subjects of both groups will have follow-up visits at 6 and 12 months and then every 12 months until 24 months after the last patient recruitment. For each group, 560 patients will be included, with an estimated total number of 1120 participants in this clinical study. Patients will be followed up until 24 months after the last enrollment.

The primary endpoint is a composite consisting of stroke, systemic embolism, cardiovascular or unexplainable death, acute coronary syndrome, coronary artery disease or periphery vascular disease requiring revascularization and major bleeding. The secondary endpoints are all-cause death, device related thrombus, minor bleeding and rehospitalization due to heart failure.

DETAILED DESCRIPTION:
The ASPIRIN LAAO trial is a prospective, multi-center, randomized, double blinded, placebo-controlled study aiming at investigating the safety of terminating the use of aspirin since the sixth month after LAAO.

Patients diagnosed with paroxysmal or persistent atrial fibrillation with an age between 18 and 90 years and have undergone LAAO will be enrolled in this study. Randomization will be performed at 6 months post-implant. The randomization program electronically assigns the patient 1:1 to either the Aspirin group or the control group. Study patients assigned to Aspirin group will receive enteric coated aspirin (100 mg/day). The control group receives placebo. After the randomization, subjects of both groups will have follow-up visits at 6 and 12 months and then every 12 months until 24 months after the last patient recruitment. For each group, 560 patients will be included, with an estimated total number of 1120 participants in this clinical study. Patients will be followed up until 24 months after the last enrollment.

The primary endpoint is a composite consisting of stroke, systemic embolism, cardiovascular or unexplainable death, acute coronary syndrome, coronary artery disease or periphery vascular disease requiring revascularization and major bleeding. The secondary endpoints are all-cause death, device related thrombus, minor bleeding and rehospitalization due to heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 90 years
* Paroxysmal, persistent, long-standing persistent or permanent nonvalvular AF
* Have already had a Watchman LAAO device implanted 6 months ago

Exclusion Criteria:

Clinical Exclusion Criteria

* Long-term aspirin therapy required
* Including coronary artery disease, symptomatic carotid disease, prior myocardial infarction, strokes or systemic embolism, etc
* Contraindicated for aspirin therapy
* Including active peptic ulcer, thrombocytopenia or anemia, etc.
* Uncontrolled malignant tumor
* Abnormal liver, renal or coagulation function
* Pregnant or pregnancy is planned during the course of the investigation
* Terminal illness with life expectancy <1 year
* Enrolled in another IDE or IND investigation of a cardiovascular device or an investigational drug

TEE Exclusion Criteria*

* Peri-device leak >5mm
* Device-related thrombus
* Other intracardiac thrombus

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 1120 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with stroke | 24 months after the date of randomization.
  A stroke is a medical condition in which poor blood flow to the brain results in cell death. There are two main types of stroke: ischemic, due to lack of blood flow, and hemorrhagic, due to bleeding. They result in part of the brain not functioning properly. Signs and symptoms of a stroke may include an inability to move or feel on one side of the body, problems understanding or speaking, dizziness, or loss of vision to one side. If symptoms last less than one or two hours it is known as a transient ischemic attack (TIA) or mini-stroke. A hemorrhagic stroke may also be associated with a severe headache. The symptoms of a stroke can be permanent. Brain computed tomography or MRI may help diagnose stroke.
Number of participants with systemic embolism | 24 months after the date of randomization.
  An embolism is the lodging of an embolus, a blockage-causing piece of material, inside a blood vessel. The embolus is usually a blood clot (thrombus). An embolism can cause partial or total blockage of blood flow in the affected vessel.
  An embolism in which the embolus is a piece of thrombus is called a thromboembolism.
  An embolism is usually a pathological event, i.e., accompanying illness or injury. Sometimes it is created intentionally for a therapeutic reason, such as to stop bleeding or to kill a cancerous tumor by stopping its blood supply.
  Embolism can be classified as to where it enters the circulation either in arteries or in veins. Arterial embolism are those that follow and, if not dissolved on the way, lodge in a more distal part of the systemic circulation.
Number of participants with cardiovascular/unexplained death | 24 months after the date of randomization.
  Cardiovascular deaths refer to deaths due to heart dysfunction, injury of cardiac structure, coronary artery diseases and lethal arrhythmias or sudden death that cannot be explain. Cardiovascular deaths can be diagnosed with clinical symptoms or from the results of diagnostic examinations.
Number of participants with major bleedings | 24 months after the date of randomization.
  Major bleedings refer to the heavy bleedings of the mains organs of the body, usually include intracranial bleeding and gastrointestinal bleeding et al.. Brain computed tomography and gastrointestinal endoscope are the common approaches for diagnosing major bleedings.
Number of participants with acute coronary syndrome | 24 months after the date of randomization.
  Acute coronary syndrome is a syndrome (set of signs and symptoms) due to decreased blood flow in the coronary arteries such that part of the heart muscle is unable to function properly or dies. The most common symptom is chest pain, often radiating to the left shoulder or angle of the jaw, crushing, central and associated with nausea and sweating. Many people with acute coronary syndromes present with symptoms other than chest pain, particularly, women, older patients, and patients with diabetes mellitus.
  Acute coronary syndrome is commonly associated with three clinical manifestations, named according to the appearance of the electrocardiogram (ECG): ST elevation myocardial infarction (STEMI, 30%), non-ST elevation myocardial infarction (NSTEMI, 25%), or unstable angina (38%). There can be some variation as to which forms of myocardial infarction (MI) are classified under acute coronary syndrome.
Number of participants with coronary or periphery artery disease requiring revascularization | 24 months after the date of randomization.
  Conronary or periphery artery diseases, regardless stable or not, need revascularization by stent which require long-term aspirin therapy

SECONDARY OUTCOMES:
Number of participants with device-related thrombus | 24 months after the date of randomization.
  This refers to the thrombus that is related to the implantation of the device for left atrial appendage closure. Transesophageal echocardiography is effective in identifying and diagnosing device-related thrombus.
Number of participants with minor bleedings | 24 months after the date of randomization.
  Minor bleedings refer to the bleedings acoording to the TIMI cirteria
Number of Participants with hospitalization due to heart failure | 24 months after the date of randomization.
  Patients need to receive treatments in hospital because of occurrence of heart failure or deterioration of heart failure.
Number of participants with all-cause death | 24 months after the date of randomization.
  any cause of death

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Gang Li, Dr., Principal Investigator — Xinhua Hospital, School of Medicine, Shanghai Jiao Tong University
Locations (1):
- Xinhua Hospital, School of Medicne, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hylek EM, Go AS, Chang Y, Jensvold NG, Henault LE, Selby JV, Singer DE. Effect of intensity of oral anticoagulation on stroke severity and mortality in atrial fibrillation. N Engl J Med. 2003 Sep 11;349(11):1019-26. doi: 10.1056/NEJMoa022913. PMID 12968085
- [Result] Mac Grory B, Chang A, Atalay MK, Yaghi S. Left Atrial Appendage Thrombus and Embolic Stroke. Stroke. 2018 Sep;49(9):e286-e289. doi: 10.1161/STROKEAHA.118.022674. No abstract available. PMID 30355001
- [Result] Piccini JP, Sievert H, Patel MR. Left atrial appendage occlusion: rationale, evidence, devices, and patient selection. Eur Heart J. 2017 Mar 21;38(12):869-876. doi: 10.1093/eurheartj/ehw330. PMID 27628431
- [Result] Reddy VY, Sievert H, Halperin J, Doshi SK, Buchbinder M, Neuzil P, Huber K, Whisenant B, Kar S, Swarup V, Gordon N, Holmes D; PROTECT AF Steering Committee and Investigators. Percutaneous left atrial appendage closure vs warfarin for atrial fibrillation: a randomized clinical trial. JAMA. 2014 Nov 19;312(19):1988-98. doi: 10.1001/jama.2014.15192. PMID 25399274
- [Result] Holmes DR Jr, Kar S, Price MJ, Whisenant B, Sievert H, Doshi SK, Huber K, Reddy VY. Prospective randomized evaluation of the Watchman Left Atrial Appendage Closure device in patients with atrial fibrillation versus long-term warfarin therapy: the PREVAIL trial. J Am Coll Cardiol. 2014 Jul 8;64(1):1-12. doi: 10.1016/j.jacc.2014.04.029. PMID 24998121
- [Result] Reddy VY, Doshi SK, Kar S, Gibson DN, Price MJ, Huber K, Horton RP, Buchbinder M, Neuzil P, Gordon NT, Holmes DR Jr; PREVAIL and PROTECT AF Investigators. 5-Year Outcomes After Left Atrial Appendage Closure: From the PREVAIL and PROTECT AF Trials. J Am Coll Cardiol. 2017 Dec 19;70(24):2964-2975. doi: 10.1016/j.jacc.2017.10.021. Epub 2017 Nov 4. PMID 29103847
- [Result] Boersma LV, Schmidt B, Betts TR, Sievert H, Tamburino C, Teiger E, Pokushalov E, Kische S, Schmitz T, Stein KM, Bergmann MW; EWOLUTION investigators. Implant success and safety of left atrial appendage closure with the WATCHMAN device: peri-procedural outcomes from the EWOLUTION registry. Eur Heart J. 2016 Aug;37(31):2465-74. doi: 10.1093/eurheartj/ehv730. Epub 2016 Jan 27. PMID 26822918
- [Result] Boersma LV, Ince H, Kische S, Pokushalov E, Schmitz T, Schmidt B, Gori T, Meincke F, Protopopov AV, Betts T, Foley D, Sievert H, Mazzone P, De Potter T, Vireca E, Stein K, Bergmann MW; EWOLUTION Investigators. Efficacy and safety of left atrial appendage closure with WATCHMAN in patients with or without contraindication to oral anticoagulation: 1-Year follow-up outcome data of the EWOLUTION trial. Heart Rhythm. 2017 Sep;14(9):1302-1308. doi: 10.1016/j.hrthm.2017.05.038. Epub 2017 May 31. PMID 28577840
- [Result] Reddy VY, Mobius-Winkler S, Miller MA, Neuzil P, Schuler G, Wiebe J, Sick P, Sievert H. Left atrial appendage closure with the Watchman device in patients with a contraindication for oral anticoagulation: the ASAP study (ASA Plavix Feasibility Study With Watchman Left Atrial Appendage Closure Technology). J Am Coll Cardiol. 2013 Jun 25;61(25):2551-6. doi: 10.1016/j.jacc.2013.03.035. Epub 2013 Apr 10. PMID 23583249
- [Result] Bosche LI, Afshari F, Schone D, Ewers A, Mugge A, Gotzmann M. Initial Experience With Novel Oral Anticoagulants During the First 45 Days After Left Atrial Appendage Closure With the Watchman Device. Clin Cardiol. 2015 Dec;38(12):720-4. doi: 10.1002/clc.22478. Epub 2015 Oct 14. PMID 26467851
- [Result] Chen S, Weise FK, Chun KRJ, Schmidt B. Antithrombotic strategies after interventional left atrial appendage closure: an update. Expert Rev Cardiovasc Ther. 2018 Sep;16(9):675-678. doi: 10.1080/14779072.2018.1510316. Epub 2018 Aug 29. PMID 30095350
- [Result] ASCEND Study Collaborative Group; Bowman L, Mafham M, Wallendszus K, Stevens W, Buck G, Barton J, Murphy K, Aung T, Haynes R, Cox J, Murawska A, Young A, Lay M, Chen F, Sammons E, Waters E, Adler A, Bodansky J, Farmer A, McPherson R, Neil A, Simpson D, Peto R, Baigent C, Collins R, Parish S, Armitage J. Effects of Aspirin for Primary Prevention in Persons with Diabetes Mellitus. N Engl J Med. 2018 Oct 18;379(16):1529-1539. doi: 10.1056/NEJMoa1804988. Epub 2018 Aug 26. PMID 30146931
- [Result] McNeil JJ, Wolfe R, Woods RL, Tonkin AM, Donnan GA, Nelson MR, Reid CM, Lockery JE, Kirpach B, Storey E, Shah RC, Williamson JD, Margolis KL, Ernst ME, Abhayaratna WP, Stocks N, Fitzgerald SM, Orchard SG, Trevaks RE, Beilin LJ, Johnston CI, Ryan J, Radziszewska B, Jelinek M, Malik M, Eaton CB, Brauer D, Cloud G, Wood EM, Mahady SE, Satterfield S, Grimm R, Murray AM; ASPREE Investigator Group. Effect of Aspirin on Cardiovascular Events and Bleeding in the Healthy Elderly. N Engl J Med. 2018 Oct 18;379(16):1509-1518. doi: 10.1056/NEJMoa1805819. Epub 2018 Sep 16. PMID 30221597
- [Result] Gaziano JM, Brotons C, Coppolecchia R, Cricelli C, Darius H, Gorelick PB, Howard G, Pearson TA, Rothwell PM, Ruilope LM, Tendera M, Tognoni G; ARRIVE Executive Committee. Use of aspirin to reduce risk of initial vascular events in patients at moderate risk of cardiovascular disease (ARRIVE): a randomised, double-blind, placebo-controlled trial. Lancet. 2018 Sep 22;392(10152):1036-1046. doi: 10.1016/S0140-6736(18)31924-X. Epub 2018 Aug 26. PMID 30158069
- [Derived] Chen M, Wang Q, Sun J, Zhang PP, Li W, Mo BF, Chen TZ, Tang X, Li YG; ASPIRIN LAAO trial investigators. Double-blind, placebo-controlled randomised clinical trial to evaluate the effect of ASPIRIN discontinuation after left atrial appendage occlusion in atrial fibrillation: protocol of the ASPIRIN LAAO trial. BMJ Open. 2021 Mar 15;11(3):e044695. doi: 10.1136/bmjopen-2020-044695. PMID 33722871